CLINICAL TRIAL: NCT01737177
Title: Bendamustine, Lenalidomide and Rituximab (R2-B) Combination as a Second-Line Therapy for First Relapsed-Refractory Mantle Cell Lymphomas: A Phase II Study
Brief Title: Bendamustine/Lenalidomide/Rituximab: Combination as a Second-Line Therapy for 1st Relapsed-Refractory MCL
Acronym: R2-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL R2-B
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Mantle Cell Lymphoma
Keywords: MCL; Mantle Cell Lymphoma; RELAPSED-REFRACTORY
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bendamustine Hydrochloride; Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustina, Lenalidomide, Rituximab (Experimental): 1 arm for all patients
  Interventions: Drug: Bendamustine, Lenalidomide, Rituximab

INTERVENTIONS:
Drug: Bendamustine, Lenalidomide, Rituximab — INDUCTION PHASE (COURSE 1-4)
  * Bendamustine: 70 mg/m2 on day 2 and 3 every 28
  * Lenalidomide: 10 mg/daily on day 1 to 14 of a 28 days course
  * Rituximab: 375 mg/m2 on day 1 every 28 days; only for the first cycle in the induction phase will start on day 8
  CONSOLIDATION PHASE (courses 5-6)
  Patients in CR and PR at the end of the induction phase
  * Lenalidomide: 15 mg/daily on day 1 to 21 of a 28 days course.
  * Rituximab: 375 mg/m2 on day 1 every 28 days
  MAINTENANCE PHASE (courses 7-24)
  Patients in CR or PR at the end of the consolidation treatment with Lenalidomide until disease progression or unacceptable toxicity up to 18 months (from month 7 to month 24)
  - Lenalidomide: 15 mg/daily on day 1 to 21 of a 28 days

SUMMARY:
This is a prospective, multicenter phase II trial designed to evaluate the safety and activity of the combination of Bendamustine, Lenalidomide and Rituximab (R2-B) in patients with first relapsed/refractory mantle cell lymphoma (MCL) and the efficacy and safety of a maintenance treatment with Lenalidomide for 18 months from the end of R2-B (from month 7 to 24) for those responding to the induction.

DETAILED DESCRIPTION:
This is a phase II study, non randomized, multicenter. Patients with MCL refractory to front line therapy or in first relapse will be enrolled.

The study includes an induction phase, a consolidation phase, a maintenance phase and a follow up phase.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a diagnosis of MCL according to the WHO classification;
* Patient age is ≥ 18 years;
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2;
* Understands and voluntarily signs an informed consent form;
* Able to adhere to the study visit schedule and other protocol requirements;
* Patients treated with one prior regimen and relapsed, or refractory to front line therapy; front line consolidation with autologous stem cell transplantation is considered to be part of first line therapy;
* Patient has at least one site of measurable nodal disease at baseline ≥ 2.0 cm in the longest transverse diameter as determined by CT scan (MRI is allowed only if CT scan can not be performed). Note: Patients with bone marrow involvement are eligible;
* Adequate haematological counts: ANC > 1.5 x 109/L and platelet count > 75 x 109/L unless due to bone marrow involvement by MCL;
* Conjugated bilirubin up to 2 x ULN unless due to liver involvement by MCL;
* Alkaline phosphatase and transaminases up to 2 x ULN unless due to liver involvement by MCL;
* Creatinine clearance ≥ 30 ml/min; a dose reduction of Lenalidomide for patients with creatinine clearance ≥ 30 mL/min but < 50 mL/min is planned;
* Written informed consent was obtained from the patient prior to any study-specific screening procedures;
* Patient has the ability to swallow capsules or tablets;
* Life expectancy ≥ 6 months;
* Disease free of prior malignancies (a part MCL) with the exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast;

Exclusion Criteria:

* Patients who have received an experimental drug or used an experimental medical device within 4 weeks before the planned start of treatment. Concurrent participation in non-treatment studies is allowed, if it will not interfere with participation in this study;
* Patient has a history of CNS involvement with lymphoma;
* Patients with previous history of malignancies (a part MCL) ≤ 3 years before study accrual with the exception of currently treated basal cell and squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix;
* History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances;
* Patient has any other concurrent severe and/or uncontrolled medical condition(s) (e.g., uncontrolled diabetes mellitus, active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol;
* Creatinine clearance < 30 ml/min;
* Patient has a known history of HIV seropositivity;
* Patient has active HBV hepatitis. The following categories of HBV positive patients but with non evidence of active hepatitis may be considered for the study and treated with R2-B (see also Section 8.1.8):
* patient is HBsAg + with HBV DNA < 2000 UI/ml (inactive carriers); HBV DNA > 2000 UI/ml is criteria of exclusion;
* patient is HBsAg - HBsAb +;
* patient is HBsAg - but HBcAb +
* Patients with HCV active hepatitis are excluded from the study. Patient with no evidence of active hepatitis and/or advanced chronic liver disease according to liver biopsy or fibro-scan evaluation may be included into the study
* Patients have received previous treatment with either Bendamustine and/or Lenalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-07-31 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Complete Response (CR) rate | At the end of the consolidation phase (6 months)
  Proportion of CR according to the Cheson2007 response criteria
Maintenance Progression Free Survival (maPFS) | 36 months
  maPFS will be defined in the maintenance cohort as the time between the date of CR/PR and the date of disease progression or death from any cause.

SECONDARY OUTCOMES:
Toxicity | 24 months
  Incidence of grade 3 or higher Toxicity measured by CTCAE v.4 during induction and maintenance therapy
Overall Response Rate (ORR) | at the end of the consolidation phase (6 months)
  ORR at the end of the consolidation treatment is defined as Complete Response(CR) or Partial Response according to the Cheson 2007 response criteria
Progression Free Survival (PFS) in all patients | 42 months
  PFS will be measured from the day of enrolment and of disease progression or death from any cause
Overall Survival (OS) | 36 months
  OS will be defined as the date of enrolment and the date of recurrence/disease progression or death from any cause
Molecular response rate | 24 months
  rate of conversion to molecular remission measured by PCR
Molecular relapse rate during study period | 42 months
  rate of conversion to molecular relapse measured by PCR
Disease kinetics of minimal residual disease (MRD) during study period | up to 42 months
  measured by real time PCR in the bone marrow and peripheral blood
Cumulative incidence of second primary malignancies | up to 42 months
  incidence of any second primary malignancies (haematological and not haematological) diagnosed after the conclusion of induction phase
To evaluate the possible relationship between Cereblon expression and response to therapy | 6 months
  Possible relationship between Cereblon expression and response to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zaja, M.D., Principal Investigator — Clinica Ematologica - Udine - Italy
Locations (43):
- Italy (43):
  - UOC Ematologia Trani, Trani, Barletta-Andria-Trani (BT)
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori IRST Meldola, Meldola, Forlì Cesena
  - Ematologia Istituto Clinico Humanitas, Rozzano, Milano
  - Centro di riferimento Oncologico CRO Aviano, Aviano, Pordenone
  - IRCCS-Centro di Riferimento Oncologico UO di Ematologia e Trapianto Cellule Staminali, Rionero in Vulture, Potenza
  - Medicina Interna 2 ad indirizzo Ematologico AOU San Luigi Gonzaga, Orbassano, Torino
  - SC Ematologia AO SS. Antonio e Biagio e C. Arrigo, Alessandria
  - Clinica di Ematologia AOU Umberto I Ospedali Riuniti, Ancona
  - SC Ematologia Spedali Civili, Brescia
  - Ematologia Ospedale Cardarelli ASREM, Campobasso
  - Oncoematologia Ospedale SS. Anna e Sebastiano, Caserta
  - UOC Ematologia Osp. Garibaldi Nesima, Catania
  - Azienda Ospedaliera Pugliese Ciaccio Dipartimento oncoematologico, Catanzaro
  - Clinica Ematologica AOU San Martino, Genova
  - Ematologia AOU S. Martino - IST, Genova
  - UOC Ematologia Universitaria Polo Pontino Sapienza, Latina
  - SC Ematologia Azienda Ospedali Riuniti Papardo Piemonte, Messina
  - UOC Ematologia Policlinico Universitario AOU G. Martino, Messina
  - SC Ematologia - Trapianto di midollo osseo Fond. IRCCS Istituto Nazionale Tumori, Milan
  - SC Ematologia AO Niguarda Cà Granda, Milan
  - SCDU Ematologia - Università del Piemonte Orientale, Novara
  - Divisione di Ematologia, Azienda Ospedali Riuniti Villa Sofia Cervello, Palermo
  - U.O. Complessa di Ematologia Ospedale di Parma, Parma
  - Ematologia Policlinico San Matteo, Pavia
  - Unità Ematologia Ospedale Civile di Piacenza, Piacenza
  - UO Ematologia Az Ospedaliera Pisana Ospedale "S.Chiara", Pisa
  - UO Ematologia Ospedale Santa Maria delle Croci, Ravenna
  - Divisione di Ematologia AO Bianchi Melacrino Morelli, Reggio Calabria
  - SC Ematologia AO Santa Maria Nuova IRCCS, Reggio Emilia
  - UO Oncoematologia ospedale degli Infermi, Rimini
  - Ematologia Ospedale San Eugenio, Roma
  - UOC Ematologia e Trapianto Istituto Regina Elena (IFO), Roma
  - Ematologia Ospedale S.Camillo Forlanini, Roma
  - Ematologia Università La Sapienza, Roma
  - UOC Ematologia AO San Giovanni Addolorata, Roma
  - Ematologia e Trapianti A.O. San Giovanni di DIO e Ruggi D'Aragona, Salerno
  - Ematologia Ospedale SG Moscati, Taranto
  - SC Oncoematologia con autotrapianto AO Santa Maria, Terni
  - SC Ematologia - AO Città della Salute e della Scienza, Torino
  - SC Ematologia U - AO Città della Salute e della Scienza, Torino
  - Clinica Ematologica ASUI Integrata di Udine, Udine
  - Oncologia Medica Varese Ospedale di Circolo e Fondazione Macchi, Varese
  - UO Ematologia Ospedale di Circolo e Fondazione Macchi, Varese